CLINICAL TRIAL: NCT07087067
Title: Early Initiation of Low-Dose Aspirin for the Prevention of Preeclampsia in High-Risk Pregnancies.
Brief Title: Aspirin Role for Preventing Clinical Risks Related to High Risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galala University (Other)
Responsible Party: Principal Investigator, Eman Hamed, Lecturer of Clinical Pharmacy, Galala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0230201
Record Dates: First submitted 2025-06-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Preeclampsia; Pregnancy
Keywords: Preeclampsia; Pregnancy; Aspirin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: 2 groups at same time
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Control (pregnant patient but not receiving Aspirin)
- Aspirin (Experimental): Receiving low dose Aspirin
  Interventions: Drug: Aspirin 75 mg

INTERVENTIONS:
Drug: Aspirin 75 mg — patients received aspirin 75 mg daily prior to 12 weeks gestation
  Arms: Aspirin

SUMMARY:
Preeclampsia and its related consequences significantly contribute to maternal and neonatal morbidity and mortality, particularly in high-risk pregnancies. Low-dose aspirin has shown promise in reducing these risks, particularly when initiated early in gestation. This study evaluated the effectiveness of 75 mg aspirin, started before 12 weeks of gestation, in reducing adverse pregnancy outcomes among high-risk pregnant women.

A randomized controlled trial was undertaken with high-risk pregnant women. Pregnant women were randomized in a 1:1 ratio to receive 75 mg of aspirin or a control daily from enrollment (<12 weeks of gestation) until 36 weeks of delivery. High-risk status was defined by established clinical criteria. The incidence of preeclampsia was the primary outcome. The researchers considered preterm birth, fetal growth restriction (FGR), perinatal mortality, neonatal intensive care unit (NICU) admission, gestational hypertension, neonatal morbidity, and postpartum hemorrhage as secondary outcomes. The outcomes were compared using Fisher's exact test, chi-square, and two-sample z-tests.

Initiation of 75 mg of low-dose aspirin early in high-risk pregnancies significantly reduced preeclampsia and several adverse neonatal outcomes without increasing maternal risk. These findings support the early start of low-dose aspirin as a safe and effective strategy for preeclampsia prevention in high-risk women.

DETAILED DESCRIPTION:
Preeclampsia continues to be one of the most severe complications of pregnancy, substantially contributing to maternal and perinatal morbidity and mortality on a global scale. It is a multisystem hypertensive disorder that frequently presents with proteinuria or symptoms of maternal organ dysfunction and typically manifests after 20 weeks of gestation. Globally, preeclampsia affects between 3% and 8% of pregnant women, with higher rates reported in resource-limited settings. Its pathogenesis is complex and multifactorial, with growing evidence pointing toward abnormal placental development and impaired spiral artery remodeling during early gestation as initiating events. This aberrant placentation leads to uteroplacental ischemia, systemic endothelial dysfunction, oxidative stress, and an amplified inflammatory response, resulting in the clinical condition of preeclampsia.

This study aimed to assess the efficacy of low-dose aspirin (75 mg daily), commenced before 12 weeks of gestation, in decreasing the occurrence of preeclampsia. and other adverse pregnancy outcomes among women with clearly defined high-risk characteristics. In contrast to prior studies with broader inclusion criteria, this trial sought to isolate the impact of aspirin in a carefully selected cohort of women at elevated risk, utilizing a randomized controlled design. 13-15 Our secondary objectives included evaluating the effects of aspirin on fetal growth restriction, neonatal morbidity, perinatal death, preterm birth, and maternal complications such as postpartum hemorrhage and gestational hypertension.

This study is a randomized controlled trial conducted between [May 2023] and [May 2025]. The trial aimed to see if starting low-dose aspirin (75 mg) early can help reduce the chances of preeclampsia and related problems for mothers and babies in pregnant women who are at high risk. This study was approved by the Ethical Committee of the Faculty of Medicine, Beni-Suef University, with approval number REC/012/005752.

Inclusion Criteria

Pregnant women were considered according to the subsequent criteria:

* Age ≥ 18 years.
* Singleton or multifetal pregnant women.
* Gestational age less than 12 weeks at the time of randomization, confirmed by first-trimester ultrasound.
* Having at least one of the major risk factors listed above.
* Being willing and able to give informed consent and follow trial processes. Exclusion Criteria

Exclusion criteria were strictly applied to reduce confounding and ensure participants' safety:

* Current or prior use of aspirin or other antiplatelet/anticoagulant therapy during the current pregnancy.
* Known hypersensitivity to aspirin.
* Peptic ulcer history, gastrointestinal bleeding, or coagulopathy.
* Platelet count <100,000/μL or known bleeding disorders.
* Severe hepatic or renal dysfunction (CKD stage IV or above).
* Known major fetal anomaly or chromosomal abnormality.
* Participation in another clinical trial that could affect outcomes. Randomization Eligible pregnant women were randomized in a 1:1 ratio to take either 75 mg of aspirin or to be assigned to the control group, commencing before 12 weeks of gestation and continuing until 36 weeks of delivery, whichever happened first. The randomization sequence was computer-generated using variable block sizes and stratified by parity (nulliparous vs. multiparous). The allocation was covered within consecutively numbered opaque envelopes Intervention The intervention group was administered a daily oral dosage of 75 mg of enteric-coated aspirin, while the control group did not receive aspirin. Medication adherence was assessed at each antenatal visit through patient diaries and tablet counts. In addition, bleeding manifestations were assessed on each visit.

Follow-up and Data Collection Participants were followed at routine antenatal care intervals until delivery. Demographic data and baseline clinical characteristics were collected at enrollment. Outcomes were prospectively recorded through standardized forms completed by trained research personnel. Delivery details and neonatal outcomes were confirmed via hospital records.

Outcome Measures Primary Outcome The American College of Obstetricians and Gynecologists (ACOG) defines preeclampsia as the following: after 20 weeks of gestation, the presence of proteinuria (≥300 mg/24 h, protein/creatinine ratio ≥0.3, or dipstick ≥1+) or indicators of maternal organ dysfunction, and new-onset hypertension (≥140/90 mmHg on two occasions at least 4 hours apart). 11, 12 Secondary Outcomes

* Preterm birth: Delivery occurring prior to 37 weeks of gestation.
* Fetal growth restriction (FGR): Birth weight under the 10th percentile for gestational age based on standardized charts.
* Perinatal death: Stillbirth at ≥20 weeks of gestation or neonatal death within 7 days of birth.
* Neonatal intensive care unit admission (NICU).
* Composite neonatal morbidity: Presence of at least one of the following-intraventricular hemorrhage (IVH), respiratory distress syndrome (RDS), hypoxic-ischemic encephalopathy (HIE), sepsis, or necrotizing enterocolitis (NEC).
* Gestational hypertension: New-onset hypertension without proteinuria or systemic findings.
* Postpartum hemorrhage (PPH) refers to the need for a blood transfusion, which occurs when there is an estimated blood loss of 500 mL or more following a vaginal delivery, 1000 mL or more following a cesarean delivery, or both.

  39 of 126 pregnant women were excluded; twenty-seven subjects didn't meet the inclusion criteria during the study enrollment, seven declined the study, four missed the follow-up, and one withdrew from the study. All 87 patients completed the randomized study: 45 in the aspirin group and 42 in the control group, as shown in Figure 1. All 87 pregnant women were included in the final analysis. Baseline demographic and clinical characteristics were well-balanced between groups. The mean maternal age was 31.4 ± 6.3 years in the aspirin group and 33.2 ± 5.9 years in the control group. Rates of chronic hypertension, pregestational diabetes, autoimmune disease, and prior preeclampsia were similar across groups, with no statistically significant differences (p > 0.05).

ELIGIBILITY:
Inclusion Criteria

Pregnant women were considered according to the subsequent criteria:

* Age ≥18 years.
* These criteria applied to both singleton and multifetal pregnant women.
* The gestational age was less than 12 weeks at the time of randomization, confirmed by a first-trimester ultrasound.
* Each participant must possess at least one of the major risk factors mentioned above.
* Being willing and able to give informed consent and follow trial processes. Exclusion Criteria

Exclusion criteria were strictly applied to reduce confounding and ensure participants' safety:

* Current or prior use of aspirin or other antiplatelet/anticoagulant therapy during the current pregnancy.
* Known hypersensitivity to aspirin.
* Peptic ulcer history, gastrointestinal bleeding, or coagulopathy.
* A platelet count of less than 100,000/μL or the presence of known bleeding disorders is a concern.
* Severe hepatic or renal dysfunction (CKD stage IV or above).
* Known major fetal anomaly or chromosomal abnormality.
* Engaging in a different clinical trial could potentially impact the results.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant females
Enrollment: 87 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
preeclampsia occurance | till end of pregnancy from week 12 to delivery
  preeclampsia occurance in high risk pregnancy in both groups

SECONDARY OUTCOMES:
Preterm birth | through study completion, an average of 1 year
  Delivery occurring prior to 37 weeks of gestation.
Fetal growth restriction (FGR): | through study completion, an average of 1 year
  Birth weight under the 10th percentile for gestational age based on standardized charts.
Perinatal death: | at ≥20 weeks of gestation or neonatal death within 7 days of birth.
  Stillbirth at ≥20 weeks of gestation or neonatal death within 7 days of birth.
Neonatal intensive care unit admission (NICU). | delivery day
  Neonatal intensive care unit admission after birth.
Composite neonatal morbidity | through study completion, an average of 1 year
  Presence of at least one of the following-intraventricular hemorrhage (IVH), respiratory distress syndrome (RDS), hypoxic-ischemic encephalopathy (HIE), sepsis, or necrotizing enterocolitis (NEC).
Gestational hypertension | through study completion, an average of 1 year
  New-onset hypertension without proteinuria or systemic findings.
Postpartum hemorrhage (PPH) | after delivery directly
  refers to the need for a blood transfusion, an estimated blood loss of 500 mL or more following a vaginal delivery or 1000 mL or more following a cesarean delivery, or both.

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Hamed, Suez, Suiz, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alsulami FT, Hamed EM. Early initiation of low-dose aspirin for the prevention of pre-eclampsia in high-risk pregnancies. Sci Rep. 2026 Jan 13;16(1):1761. doi: 10.1038/s41598-025-28078-3. PMID 41530193